CLINICAL TRIAL: NCT01372371
Title: Effects of Applying Powdered Prophylactics Verses Intravenous Antibiotics Only on Post-operative Infection Rate
Brief Title: Efficacy of Local Powder Prophylactics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ganga Hospital (Other)
Responsible Party: Dr. S. Rajasekaran, Ph.D., Ganga Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1119-9648
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Infection
Keywords: Vancomycin, Gentamycin; Local Powder Antibiotic's Efficacy in Controlling Post Surgical Infection
MeSH Terms: conditions — Infections | interventions — Vancomycin; Gentamicins; Cefuroxime

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vancomycin (Active Comparator)
  Interventions: Biological: Vancomycin
- Vancomycin and Gentamycin (Active Comparator)
  Interventions: Biological: Vancomycin and Gentamycin
- Intravenous Antibiotic (Active Comparator)
  Interventions: Biological: Cefuroxime

INTERVENTIONS:
Biological: Vancomycin — 1 pre-operative dose of intravenous Cefuroxime (1.5 gm) and 2 post-operative doses of Cefuroxime (750 mg) + 500 mg of vancomycin instilled on surgical site before closure
  Arms: Vancomycin
Biological: Vancomycin and Gentamycin — 1 pre-operative dose of intravenous Cefuroxime (1.5 gm) and 2 post-operative doses of Cefuroxime (750 mg) and 500 mg of vancomycin powder on surgical site before closure with gentamycin bone cement for joint replacement cases.
  Arms: Vancomycin and Gentamycin
Biological: Cefuroxime — 1 pre-operative dose of Cefuroxime (1.5 gm) and 2 post-operative doses of Cefuroxime (750 mg)
  Arms: Intravenous Antibiotic

SUMMARY:
Hypothesis: Directly applying antibiotic powder onto the site of surgery along with perioperative intravenous antibiotics, before closing the wound, is more effective than intravenously applied perioperative antibiotics alone in controlling post-operative wound infection. The investigators also think powders that control both gram positive and gram negative bacteria are more beneficial.

DETAILED DESCRIPTION:
1. Subjects will be divided into three groups based on the procedure used for the application of antibiotics

   1. No local antibiotics (control group): In this group, individuals will be subjected to peri-operative intravenous* antibiotics only
   2. Gram positive antibiotic: In this group, gram positive (powdered vancomycin)+ will be applied to the site of surgery, before closure of the wound, along with peri-operative intravenous antibiotics*
   3. Gram positive and gram negative: In this group, gram positive (powdered vancomycin) will be instilled on the site of surgery, before closing the wound, and gram negative antibiotic (gentamycin mixed with bone cement)+ will be used, along with peri-operative intravenous antibiotics* (only in cases of implant fixation).

      * Intravenous antibiotic dosage: 1 pre-operative dose of Cefuroxime 1.5 gm and 2 post-operative doses of Cefuroxime 750 mg.

        * Vancomycin and Gentamycin dosage: 500 mg of vancomycin powder will be used and in group 'c' gentamycin mixed with bone cement will be used along with vancomycin powder.
2. Sample size: Based on, finding at least 4% difference between the proportions of infections found in control (generally 5%, 4% in case of joint replacement) and case groups (1%) (proportions were assumed from literature and our institute records), a sample size of minimum 285 in each group (424 for joint replacement cases) will be considered for the observation to be significant at an alpha level of 0.05. This will give the study a minimum power of 80%.

   Spine cases: Control = 143, Gram-P = 143; Trauma cases: Control = 143, Gram-P = 143; Joint replacement cases: Control = 424, Gram-P = 424, Gram-P+Gram-N = 424; Total = 1844; Where Control - Cases with intravenous antibiotic dose; Gram-P - Cases with intravenous antibiotic + local antibiotic (Vancomycin, acts against gram positive bacteria); Gram-N - Cases with intravenous antibiotic + local antibiotic (Vancomycin, acts against gram positive bacteria) + local Gentamycin cement (acts against gram negative bacteria).
3. Procedure: Sampling will be based on stratified procedure. The total sample will be divided into categories based on the type of surgery, which are spine, trauma and joint replacement. Subjects within each category will be randomly selected for the three antibiotic treatments. For this study, we will use computer software to generate restricted randomization to achieve balance between groups in size. Within this restricted randomization, single block random size will be used to ensure randomization within each group.

   While joint surgery category will have all the three groups of cases (a, b and c), spine and trauma surgery category will have only two groups (a and b). Surgeries will be performed accordingly i.e. control group individuals will undergo mandated hospital policy requirements + perioperative intravenous antibiotic treatment and cases will undergo mandated hospital policy requirements + powdered vancomycin, or both vancomycin, just before the closure of the wound, and gentamycin as a mix with bone cement. Patients who exhibit both superficial and deep wood infection will be considered as infected and accounted for statistical analysis.
4. Analysis: Our main parameter of comparison is infection percentage among control and cases. Various factors like duration of surgery, tourniquet time, prior infections, blood transfusion, haemoglobin count, comorbidities, etc, will be considered while analysing for infection percentage. Infection proportions will be compared between different groups at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All joint replacement patients
* All non infected spine patients
* Hemiarthroplasty, All upper limb plating of closed fractures

Exclusion Criteria:

* Open injuries in trauma
* Revision joint replacement surgeries
* Patients with suspicion of existing infection

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1844 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Infection percent after surgery | Within one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rajasekaran Shanmuganathan, Ph.D., Principal Investigator — Ganga Hospital
Locations (1):
- Ganga Hospital, Orthopaedics Department, Coimbatore, Tamil Nadu, India